CLINICAL TRIAL: NCT06886698
Title: Arterial Spin Label Assessment of Cerebral Blood Flow in Anesthetized Children
Brief Title: MRI Assesment of Cerebral Blood Flow in Anesthetized Children
Acronym: BAMBI
Status: Not yet recruiting | Type: Observational
Sponsor: Karolinska Institutet (Other)
Collaborators: Karolinska University Hospital (Other)
Responsible Party: Principal Investigator, Jacob Karlsson, PI, Karolinska Institutet
Other Study IDs: K 2025-0337; Region Stockholm (Other: Region Stockholm)
Record Dates: First submitted 2025-03-13; First posted 2025-03-20 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Blood Flow; Cerebral Oxygenation; Blood Pressure
Keywords: anesthesia; bloodflow; brain; children

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- pediatric MRI: Patients scheduled for brain MRI under anesthesia, aged 6 months to 12 years.

SUMMARY:
Children undergoing magnetic resonance imaging (MRI) of the brain often need to be sedated to complete the examination, as it is difficult to remain still for a long period, which is required to obtain usable images. During sedation, most patients typically experience a drop in blood pressure, including children. Maintaining an adequate blood pressure under anesthesia is important, as blood pressure is routinely used as a measure to ensure sufficient blood circulation to the body's organs, including the brain. Ensuring adequate blood flow to the brain is one of the cornerstones of all anesthesia, including in children. Therefore, low blood pressure during anesthesia is often treated with standardized interventions, such as blood pressure-raising interventions. These treatments generally restore blood pressure to normal, but how this affects blood flow to the brain in children is not fully known.

With the help of modern MRI technology (so-called Arterial Spin Labeling, ASL), blood flow in the brain can be measured quickly and completely safely with high precision.

In similar situations with adult patients, it has been observed that while blood pressure-raising interventions successfully normalize low blood pressure, MRI scans show that blood flow to the brain paradoxically decreases despite the increase in blood pressure. It is believed that this may be due to the brain's blood vessels constricting.

The investigators now wish to examine this relationship in sedated children undergoing planned brain MRI for certain diagnoses. The investigators hypothesis is that standardized measures intended to raise blood pressure (i.e., the routine treatment used regardless of whether a patient participates in the study or not) normalizes low blood pressure (when deemed necessary to treat according to routine) but does not necessarily lead to improved blood flow to the brain.

Primary research question: How does routine treatment of low blood pressure affect cerebral blood flow in sedated children?

DETAILED DESCRIPTION:
Patients undergoing sedation for brain MRI will be identified based on the surgical schedule . If no exclusion criteria are met, the child will be eligible for inclusion in the study, and both the child and their guardians will be informed, with consent requested and obtained.

Basic data regarding the patient's health status, age, sex, and weight will be collected and stored on a dedicated research computer.

The anesthesia procedure for MRI examinations routinely involves measuring blood pressure before administering premedication. A peripheral venous catheter (PVC) is then placed, after which the child is sedated with a propofol infusion (an anesthetic drug). Oxygen is routinely provided via nasal cannula. Standard monitoring includes heart rate, blood pressure, and blood oxygen saturation. All study participants will be prepared, sedated, and monitored according to this standard procedure, exactly as would be done regardless of whether they participate in the study or not.

Once the child is placed in the MRI scanner, the examination proceeds as per routine. Blood pressure is measured every five minutes. As soon as the mean arterial pressure (MAP) drops by more than 20% from baseline (i.e., the blood pressure measured when the patient was awake), brain blood flow measurement using an ASL sequence in the MRI machine will begin. ASL, or Arterial Spin Labeling, is a safe MRI technique for measuring cerebral blood flow without the need for contrast injection. This method magnetically "labels" the blood and then tracks its movement into the brain, providing valuable information about cerebral perfusion. ASL is already routinely used in children undergoing MRI for conditions such as epilepsy, brain tumors, and headaches.

The ASL sequence will be initiated immediately upon detecting the blood pressure drop. Subsequently, blood pressure will be managed according to clinical routine (this management will be performed regardless of study participation), and brain blood flow will be recorded during the ASL sequence. Clinical routine management primarily involves administering intravenous blood pressure-raising medications. The ASL sequence itself takes approximately 12 minutes. Once the study protocol is completed, the MRI examination and anesthesia/monitoring will continue as per routine until completion.

Data collected from the ASL scans will then be processed using specialized software for further analysis. ASL recording will begin upon detecting a >20% drop in blood pressure, after which blood pressure will be treated according to routine. Normally, no pre-prepared blood pressure treatment is available, meaning it must be prepared at the time (e.g., blood pressure-raising medication). This preparation is estimated to take approximately 3 minutes, so the additional 12-minute sequence effectively extends the MRI duration by about (12-3) = 9 minutes (practically, this is expected to add around 10-15 extra minutes). In context, this additional time is negligible for the patient, as time windows of 10-15 minutes are common during MRI, for example, when waiting for image interpretation or adding new sequences (such as ASL, which is sometimes included for additional information, regardless of study participation).

The study will not result in an increased number of visits for research participants

ELIGIBILITY:
Inclusion Criteria:

* children aged 6 months to 12 years
* Planned to undergo MRI brain
* Exclusion Criteria:
* known brain tumor
* vascular malformation in the brain
* hydrocephalus

Ages: 6 Months to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Patients scheduled for brain MRI under anesthesia, aged 6 months to 12 years
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2025-04-15 (Estimated); Primary Completion 2026-04-15 (Estimated); Study Completion 2026-09-15 (Estimated)

PRIMARY OUTCOMES:
Changes in cerebral blood flow in response to hypotension treatment | From detection of hypotension to assessment of immediate change in cebrebral bloodflow, data reported after approximately one year
  Quantification of cerebral blood flow using Arterial Spin Labeling during hypotension and subsequently in response to standardized treatment of hypotension as per departmental standard operating procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Jacob Karlsson, MD PhD Associate Professor, Principal Investigator — Karolinska Universitets Sjukhuset
Locations (1):
- Karolinska University Hospital, Solna, Sweden

IPD SHARING:
Plan to Share IPD: Undecided